CLINICAL TRIAL: NCT05244655
Title: Early Postoperative Pain and 30-day Complications Following Major Abdominal Surgery: an Observational Study
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CORE-1
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2021-11

CONDITIONS: Infectious Complications; Postoperative Pain; Acute Pain; Postoperative Complications; Surgery--Complications
Keywords: Early postoperative pain; Infectious complications
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without painscores available during hospital stay
- Patients with painscores available during hospital stay

SUMMARY:
In this retrospective cohort study, we assess the relationship between the intensity of early postoperative pain and the risk of infectious- and non-infectious complications within 30 days after major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery under general anesthesia

Exclusion Criteria:

* younger than 18 years of age
* procedures outside the operation room
* procedures solely under regional anesthesia, i.e. no general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who underwent major abdominal surgery, mostly electively scheduled, between January 2014 and December 2020 were considered eligible for participation in our study.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Acute postoperative pain | 1 day
  Early pain following abdominal surgery POD1

SECONDARY OUTCOMES:
Infectious complications postoperative | 30 days
  within 30 days
Overall complications postoperative | 30 days
  within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bijkerk V, Jacobs LMC, Visser J, van Helden EV, Keijzer C, Helder LS, Albers KI, Warle MC. The immunomodulatory effect of sugammadex in vitro and after total hip arthroplasty : A randomised controlled pilot and retrospective cohort study. Eur J Anaesthesiol. 2025 Aug 1;42(8):676-686. doi: 10.1097/EJA.0000000000002132. Epub 2025 Feb 14. PMID 39957489